CLINICAL TRIAL: NCT04769206
Title: Enhancing Parasympathetic Activity to Improve Endothelial Dysfunction, Vascular Oxidative Stress in African Americans
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Cyndya Shibao, MD, Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202376
Record Dates: First submitted 2021-02-20; First posted 2021-02-24 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Endothelial Dysfunction
Keywords: African American; Flow-mediated dilation (FMD); Vascular Oxidative Stress
MeSH Terms: interventions — Galantamine; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Galantamine (Experimental): Galantamine 16mg/day
  - titrating: 4mg once a day for 2 weeks, titrate to 8mg once a day for 2 weeks, then 8mg twice a day for 8 more weeks
  Interventions: Drug: Galantamine
- Placebo (Placebo Comparator): placebo (micro crystalline cellulose)
  - 1 pill once daily for 4 weeks, then 2 pills daily for 8 weeks
  Interventions: Drug: Placebo
- TENS 7000 (Active Comparator): Substudy: the effect of trans-auricular vagus nerve stimulation (TaVNS) will be done by FDA-approved TENS 7000 device and during a period of enhanced vascular oxidative stress
  Interventions: Device: TENS 7000

INTERVENTIONS:
Drug: Galantamine — 4mg daily titrating up to 8mg twice a day
  Other Names: Razadyne
  Arms: Galantamine
Drug: Placebo — 1 pill a day for 4 weeks, 2 pills a day for 8 weeks
  Other Names: sugar pill
  Arms: Placebo
Device: TENS 7000 — The FDA-approved TENS 7000 device will be used for Trans-auricular vagus nerve stimulation (TaVNS) during a period of enhanced vascular oxidative stress. This device will be supplemented with ear clip electrodes. The site of the stimulation for such electrodes are the tragus or concha. The device will have built in safety controls to minimize additional risks to the subjects (as per FDA guidance on stimulators). We will use typical stimulation conditions (30 Hz, 300 µs) and amplitude dependent on perception threshold.
  Arms: TENS 7000

SUMMARY:
Specific Aim 1: To test the hypothesis that prolonged (3-month) treatment with galantamine inhibits NADPH IsoLG-protein adducts formation and improves markers of endothelial cell (EC) dysfunction in AAs.

Aim 1a: The investigators will determine if galantamine inhibits NADPH IsoLG-protein adducts formation, superoxide production, and immune cell activation compared to placebo.

For this purpose, the investigators will study peripheral blood mononuclear cell (PBMC), a critical source of systemic oxidative stress, collected from study participants.

Aim 1b: The investigators will determine if galantamine reduces intracellular Iso-LGs, ICAM-1, and 3-nitrotyrosine, a marker of vascular oxidative stress, in ECs harvested from study participants.

Specific Aim 2: To determine if prolonged (3-month) treatment with galantamine improves endothelial dysfunction as measured by vascular reactivity in AAs. The investigators will measure vascular reactivity in response to ischemia in two vascular beds: (a) in conduit arteries (brachial artery) using brachial artery diameter flow-mediated dilation (FMD), and (b) in the microvasculature (MBV) using contrast-enhanced ultrasonography in skeletal muscle.

Sub-study (optional) Will study the effect of trans-auricular vagus nerve stimulation (TaVNS) during a period of enhanced vascular oxidative stress

This proposal will study a novel mechanism that could alter the oxidative and immunogenic responses that contributes to endothelial dysfunction in AAs and will offer a potential pathway for the development of more effective therapies aimed at decreasing the progression of endothelial dysfunction to cardiovascular disease in this population.

DETAILED DESCRIPTION:
Endothelial dysfunction, a pro-thrombotic, inflammatory condition that causes impaired vascular reactivity is an early reversible step in the development of atherosclerosis and cardiovascular disease (CVD). Multiple studies consistently shown that African Americans (AAs) have impaired endothelial function compared to whites. African Americans also experience disproportionately higher CV morbidity and 20% higher mortality than whites or Hispanics. Endothelial dysfunction is caused by the overproduction of reactive oxygen species (ROS), particularly superoxide which interferes with endothelial-derived nitric oxide signaling pathways. One of the major sources of superoxide is NADPH oxidase; our previous work found that activation of NADPH oxidase contributes to vascular oxidation through the formation of highly immunogenic isolevuglandins (IsoLG-protein adducts) in peripheral mononuclear cells (PBMCs), which stimulates antigen presenting cells (APC) and inflammatory mediators. Inflammation and oxidative stress are modulated by the parasympathetic nervous system (PNS). The investigators and others found that AAs have reduced PNS activity compared with whites. Studies in animal models have shown that parasympathetic nervous stimulation with either acetylcholinesterase inhibitors or direct vagus nerve stimulation protect against oxidative stress and inflammation

There is Sub-study (optional) attached to the above main study. It is to evaluate the effect of trans-auricular vagus nerve stimulation (TaVNS) during a period of enhanced vascular oxidative stress. It is an ancillary, mechanistic, proof-of-concept study to determine if acute vagal stimulation with a Transcutaneous Electrical Nerve Stimulation device (TENS) inhibits immune cell activation and improves markers of endothelial cell dysfunction.

The investigators preliminary data in obese AA women found that stimulation of the PNS cholinergic transmission with the acetylcholinesterase inhibitor, galantamine, blocked the production of oxidative stress and inflammatory cytokines induced by lipids.

The overall goal of the current proposal is to determine if prolonged treatment with galantamine improves endothelial dysfunction and vascular oxidative stress in AAs. For this purpose, the investigators will conduct a proof-of-concept, blinded, randomized, placebo-controlled study to test the effect of 3-month treatment with galantamine (16 mg/day) on vascular oxidative stress and impaired vascular reactivity in AAs.

A total of 160 participants enrolled and will be randomized, so that we can complete 88 AAs (44 per treatment arm) in a 1:1 ratio to 8 mg p.o. twice a day (16 mg/day) of galantamine

Screening visit: After the informed consent process, subjects will undergo a history and physical examination. Other tests include EKG, collection of fasting blood samples: cell blood count, lipid profile, comprehensive metabolic panel and HbA1c.

Randomization (V1): Two antecubital IVs will be placed for EC harvesting, blood collection, and drug infusion; we will monitor continuous blood pressure and ECG throughout the study to evaluate for cardiovascular autonomic parameters. Subjects will then be challenged with an intralipid infusion to stimulate oxidative stress, and the assessment of endpoints will be performed.

After completing visit 1 procedures, and prior to being discharged, the subjects will be randomized to 8 mg p.o. twice a day (bid) (16 mg/day) galantamine or matching placebo in a 1:1 ratio using a block randomization algorithm with random block size and the assignments will be blinded to the investigator and the study subject.

Telemedicine visits: The study nurse will conduct telemedicine visits with the study subject at 1, 3 and 5 days after the initiation of the study drug to evaluate for drug's side effects.

Safety follow-up visits (V2, V3, V4): Subjects will be asked to attend three outpatient clinic visits at 2, 4 and 8 weeks that coincide with the dose-titration schedule. The first dose will be 4 mg a day for 2 weeks (visit 1, V1), then they will increase it to 8 mg a day for 2 weeks (visit 2, V2) and then 8 mg twice a day (visit 3, V3) for the remainder of the study.

Final assessment of endpoints Visit 5 (V5): The blinded medication will be administered at 7:00 AM before any procedure is performed. The subject will repeat the procedures outlined in V1.

Sub study (Optional): Mentoring in cholinergic regulation of vascular oxidation

This pilot study is an open-label, before-after design. The total sample size for Aims 1 and 2 is 12 subjects. Subjects of those completing the parent trial will meet the inclusion criteria, will return for an additional visit (V6)

Aim 1: To test the hypothesis that acute vagal stimulation with TaVNS inhibits immune cell activation. For this purpose, we will determine NADPH IsoLG-protein adducts formation, superoxide production, and immune cell activation in peripheral blood mononuclear cells (PBMC), a critical source of systemic oxidative stress, before and after lipid-induced ROS production, during continuous TaVNS. Aim 2: We will determine if acute vagus nerve stimulation with TaVNS inhibits endothelial cell dysfunction. For this purpose, we will assess intracellular Iso-LGs, ICAM-

1, and 3-nitrotyrosine, a marker of vascular oxidative stress, in harvested ECs before and after lipid-induced ROS production during continuous TaVNS.

Subjects of those completing the parent trial, will return for an additional visit (V6). This visit will be scheduled at least 4 weeks after V5 (end of parent trial) to allow wash-out of the blinded study medication and maintain the blind of the parent study. Subjects will be instrumented for TaVNS, before been challenged with an intralipid infusion to stimulate oxidative stress, and the assessment of endpoints will be performed. PBMCs will be collected before, at 2 and 4 hours after lipid infusion to assess for NADPH activation (aim 1) and will also harvest ECs before and after lipid infusion to assess for intracellular IsoLG-protein adducts, ICAM-1, and 3-nitrotyrosine in harvested ECs. ECs will be harvested using four sterile J-wires.

Primary Intervention (TaVNS) The FDA-approved TENS 7000 device for the treatment of pain will be used for TaVNS. This device will be supplemented with ear clip electrodes. The site of the stimulation for such electrodes are the tragus or concha

Specifically, the investigators will evaluate whether 3 month of galantamine treatment inhibits the activation of NADPH-IsoLG formation and the subsequent immunogenic responses in PBMCs. Furthermore, the investigators will determine if galantamine decreases markers of oxidative stress and inflammation in harvested endothelial cells (ECs) and improves vascular reactivity in the same study subjects. The planned studies will provide a comprehensive assessment of the mechanism underlying the effect of increased PNS cholinergic transmission on endothelial dysfunction.

If the investigators' hypothesis is correct, and galantamine improves endothelial dysfunction in AAs, a population with a high risk for CVD, they will discover a novel mechanism that could alter the oxidative and immunogenic responses in this population and will offer a potential pathway for the development of more effective therapies aimed at decreasing CVD.

The parent study along with the Sub study offers a novel research approach with advanced skills in using both a pharmacological intervention that enhances cholinergic activity and direct vagus nerve stimulation. These approaches could generate more effective therapies aimed at decreasing the progression of endothelial dysfunction to cardiovascular disease African Americans.

ELIGIBILITY:
Inclusion Criteria:

1. African American women and men
2. Age 18 to 60 years old
3. BMI >28

Exclusion Criteria:

1. Individuals with a history of physician diagnosed myocardial infarction, angina, heart failure, stroke, or transient ischemic attack, or who had undergone an invasive procedure for CVD (coronary artery bypass graft, angioplasty, valve replacement, pacemaker placement or other vascular surgeries)
2. Uncontrolled hypertension defined as persistent blood pressure >140/90 despite the use of anti-hypertensive agents.
3. Diabetes Mellitus type 1 or type 2, as defined by a fasting plasma glucose of 126 mg/dL or greater hemoglobin A1C (HbA1C) 6.5% or above or the use of anti-diabetic medication
4. The use of nitrates.
5. The metabolism of galantamine is primarily through the cytochrome P450 system, specifically the CYP2D6 and CYP3A4 isoenzymes. We will exclude subjects who have impaired hepatic function and/or who are currently using strong inhibitors of CYP3A4 and CYP2D6 (e.g. ketoconazole and paroxetine, respectively).
6. Pregnancy or breast-feeding. Women of child-bearing potential will be required to have undergone tubal ligation or to be using an oral contraceptive or barrier methods of birth control.
7. Post-menopausal women.
8. The use of any other central or peripheral acetylcholinesterase inhibitor (donezepil (Aricept(R)), pyridostigmine (Mestinon(R)), rivastigmine (Exelon(R)), tacrine (Cognex(R)).
9. First, second or third-degree AV block detected during the screening visit with an ECG
10. Seizures or history of seizures.
11. Current smokers defined as those who smoked a cigarette in the last 30 days.
12. History of recurrent syncope.
13. History of serious neurologic disease such as cerebral hemorrhage, stroke, or transient ischemic attack.
14. History of cardiac shunts.
15. Allergy to eggs or soy.
16. Impaired hepatic function (aspartate amino transaminase [AST] and/or alanine amino transaminase [ALT] >3.0 x upper limit of normal range)
17. Impaired renal function test (eGFR<60 mL/min/1.73m2)
18. Anemia (hematocrit <34%)
19. Ongoing substance abuse.
20. Treatment with any investigational drug in the one month preceding the study
21. Mental conditions rendering a subject unable to understand the nature, scope and possible consequences of the study
22. Inability to comply with the protocol, e.g. uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
FMD | From baseline to 3 months
  flow mediated dilation
NADPH activation in PBMC | From baseline to 3 months
  NADPH activation as measured by subunits p47phox/gp91 phox in PBMC
NADPH activation in PBMC at TaVNS stimulation | From baseline to 120 mins to 240 mins
  NADPH activation as measured by subunits p47phox/gp91 phox in PBMC.pre- and post-device stimulation measurements before( baseline) and after lipids infusion at 2 and 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Cyndya Shibao, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Chaney Johnson, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No